CLINICAL TRIAL: NCT06948136
Title: Acute Effects of THC in Older Adult
Acronym: THC-Aging
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Deepak C. D'Souza, Professor of Psychiatry, Yale University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 2000038388; 1R21DA058138-01A1 (NIH)
Record Dates: First submitted 2025-01-21; First posted 2025-04-29 (Actual); Last update posted 2025-08-18 (Actual); Status verified 2025-08

CONDITIONS: Age-related Cognitive Decline
MeSH Terms: interventions — Dronabinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Delta-9-THC Very Low Dose (Active Comparator): Active delta-9-THC administered intravenously over 20 minutes.
  Interventions: Drug: Delta-9-THC Low Dose
- Placebo (Placebo Comparator): Control: Small amount of alcohol administered intravenously (quarter teaspoon), with no delta-9-THC, over 20 minutes.
  Interventions: Drug: Placebo
- Delta-9-THC Medium Dose (Active Comparator): Active delta-9-THC administered intravenously over 20 minutes.
  Interventions: Drug: Delta-9-THC Medium Dose

INTERVENTIONS:
Drug: Delta-9-THC Low Dose — Active Delta-9-THC administered intravenously over 20 minutes.
  Arms: Delta-9-THC Very Low Dose
Drug: Placebo — Small amount of sterile ethanol (1-2 mLs), with no THC, administered intravenously over 20 minutes.
  Arms: Placebo
Drug: Delta-9-THC Medium Dose — Active Delta-9-THC administered intravenously over 20 minutes
  Arms: Delta-9-THC Medium Dose

SUMMARY:
The primary objective of this study is to determine if increasing age confers greater vulnerability to the acute A) cognitive (e.g., memory, attention, psychomotor function), B) subjective (e.g., anxiogenic and rewarding effects), and C) cardiovascular (heart rate and blood pressure), effects of THC in adults > 21 years old. The secondary aims of the study are to explore age-related acute effects of THC on electrophysiological indices of information processing (e.g., auditory steady-state response (ASSR), oddball paradigm [P300], and resting state cortical noise) and to determine age-related differences in the metabolism of THC.

ELIGIBILITY:
* Ability to provide informed consent
* No history (current or past) of unstable or serious medical, neurological or psychiatric conditions.
* High school education or greater
* No positive pregnancy test and/or lactation/ planning to nurse while in this study
* English speaking

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-06 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Rey Auditory Verbal Learning Task (RAVLT) total immediate recall | Each test day will be split into two drug administration sessions. The RAVLT will be administered approximately 25 minutes after each drug administration.
  The task consists of 5 trials, an interference list, free delayed recall, and recognition.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | -60 minutes, 20 minutes, 60 minutes, 120 minutes, 170 minutes, 210 minutes, 270 minutes, 300 minutes, 360 minutes, 420 minutes after the start of the initial THC/placebo drug infusion.
  Various feeling states will be measured using a self-reported visual analog scale of feeling states (ex: "calm and relaxed", and "tired") associated with drug administration. Subjects will be asked to score the perceived intensity of these feeling states at that moment on a 100 mm line (0 = not at all, 100 = extremely). A higher score reflects a positive response.

CONTACTS AND LOCATIONS:
Overall Officials: Deepak C D'Souza, MD, Principal Investigator — Yale University School of Medicine; VA Connecticut Healthcare System; Ashley Schnakenberg Martin, PhD, Principal Investigator — Yale University School of Medicine; VA Connecticut Healthcare System
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States